CLINICAL TRIAL: NCT03305705
Title: Double-Blind, Single-Center Interventional Trial To Evaluate The Effect Of Intravenous Iron Versus Placebo On Cerebral Dopamine Receptor Density In Non Anaemic Premenopausal Women With Low Ferritin Levels And Fatigue
Brief Title: Effect of Iron on Cerebral Dopamine Receptor Density in Non-anaemic Premenopausal Women With Low Ferritin and Fatigue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Albina Nowak, MD (Other)
Responsible Party: Sponsor-Investigator, Albina Nowak, MD, senior physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: BASEC-Nr. PB_2017-00429; KEK-ZH-Nr. 2014-0217 (Other: KEK Zurich)
Record Dates: First submitted 2017-09-19; First posted 2017-10-10 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Fatigue; Iron-deficiency
MeSH Terms: conditions — Fatigue; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will be blinded with respect to the treatment sequence. The outcome assessor (PET scan evaluator) will be blinded with respect to the participant identity and the date of the PET scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm 1 (Experimental): Patients will be treated with 0.9% sodium chloride (placebo) at Visit 1 and with iron carboxymaltose in 6 weeks at Visit 2. The patients will be blinded with respect to the treatment sequence.
  Interventions: Drug: Iron Carboxymaltose; Drug: Sodium chloride 0.9%
- Treatment Arm 2 (Experimental): Patients will be treated with 0.9% sodium chloride (placebo) at Visit 1 and with iron carboxymaltose in 6 weeks at Visit 2. The patients will be blinded with respect to the treatment sequence.
  Interventions: Drug: Iron Carboxymaltose; Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Iron Carboxymaltose — Single intravenous infusion within 20 min
  Other Names: Ferinject®
Drug: Sodium chloride 0.9% — Single intravenous infusion of 250 ml within 20 min
  Other Names: NaCl 0.9 % (serves as Placebo)

SUMMARY:
This study investigates the effect of intravenous iron substitution in non-anaemic premenopausal women with iron deficiency on:

* Changes in the cerebral Dopamine (DA) receptor density after iron substitution, shown by brain PET
* Reduction of fatigue and other neuropsychological symptoms after iron supplementation

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects, Age > 18 years, premenopausal, regularly menstruating
* BMI 18-25 kg/m2
* Serum ferritin level < 15 μg/ml, Hb > 120 g/L
* Adequate contraception during the study period
* Fatigue determined as 2 or more points in the basic questionnaire for fatigue
* Informed consent

Exclusion Criteria:

* Day-night shift work
* 11 or more points in the BDI
* No psychiatric disease (as assessed by neuropsychiatric assessment)
* 15 or more points in the ISI
* Known hypersensitivity to iron carboxymaltose, iron sucrose or iron sulfate
* Intake of iron preparations during the last 8 weeks before the start of the trial protocol
* Pregnancy or lactation
* Any cardiovascular or pulmonary disease
* Acute or chronic infection/inflammation or malignancy
* Other obvious physical or psychiatric causes for fatigue (known mental disorders, e.g. depression)
* Chronic intake of concurrent medication (especially antipsychotic drugs), except oral contraceptives. Sporadic intake of NSAID or paracetamol, e.g. in the case of a common cold or sporadic headaches is allowed.
* CRP > 10 mg/L
* TSH out of normal range
* Any concurrent medical condition(s) that, in the view of the investigator, would prevent compliance or participation or jeopardize the health of the patients.
* Participation in any other therapeutic trial within the previous month
* Known History of HIV/HBV/HCV

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-23 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Dopamine (DA) receptor density | 6 weeks
  Changes in the cerebral Dopamine (DA) receptor density determined by brain PET with the 11C-Raclopride tracer

SECONDARY OUTCOMES:
Fatigue | 6 weeks
  Reduction of fatigue after iron supplementation determined by Fatigue Assessment Scale (FAS)
Fatigue | 6 weeks
  Reduction of fatigue after iron supplementation determined by "Würzburger Erschöpfungs-Inventar bei Multipler Sklerose" (WEIMuS, in German) questionaire
Neuropsychological symptoms | 6 weeks
  Reduction of neuropsychological symptoms after iron supplementation determined by neuropsychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Albina Nowak, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No